CLINICAL TRIAL: NCT01924221
Title: Study of Reverse Electrical Remodeling of Native Conduction in Cardiac Resynchronization Therapy
Brief Title: Reverse Electrical Remodeling of Native Conduction in Cardiac Resynchronization Therapy
Acronym: RER-CRT
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00065477
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Heart Failure; Patients Undergoing CRT-D Device Implantation
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CRT: Patients with implanted cardiac resynchronization therapy defibrillator

SUMMARY:
Cardiac resynchronization therapy with pacemaker alone, or in combination with a cardioverter-defibrillator, prolongs life and decreases risk of heart failure exacerbation in patients with low ejection fraction and wide QRS. Some patients achieve decrease in QRS duration 6 months after cardiac resynchronization therapy. Such phenomenon is called reverse electrical remodeling of native conduction. Retrospective analysis showed that reverse electrical remodeling of the native conduction after at least 6 months of CRT is associated with decreased rate of ventricular arrhythmias and better survival. This study is designed to study reverse electrical remodeling prospectively.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing implantation of a CRT-D

Exclusion Criteria:

* age < 18 y
* pregnancy or planned pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Failure Patients undergoing implantation of cardiac resynchronization therapy defibrillator
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
correlation between electrical and mechanical remodeling | 6 months after CRT implantation
  correlation between electrical and mechanical measures of dyssynchrony

CONTACTS AND LOCATIONS:
Overall Officials: Larisa Tereshchenko, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States